CLINICAL TRIAL: NCT03832244
Title: The Role of Sub-mental Ultrasonography in Diagnosing Obstructive Sleep Apnea and Its Correlation With Subjective Scales
Status: Completed | Type: Observational
Sponsor: Bartin State Hospital (Other Government)
Responsible Party: Principal Investigator, Ozgeyagcioglu Yassa, Principal Investigator, Bartin State Hospital
Other Study IDs: BartinUyku
Record Dates: First submitted 2019-02-03; First posted 2019-02-06 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Obstructive Sleep Apnea; Diagnostic Imaging; Ultrasound
Keywords: sub-mental ultrasonography; obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Simple snoring: Patients undergoing to Sub-mental ultrasonography with Normal sleep: Fewer than 5 events per hour measured in over-night polysomnography
  Interventions: Diagnostic Test: Sub-mental ultrasonography
- Mild OSA: Patients undergoing to Sub-mental ultrasonography with Mild sleep apnea: 5 to 14 events per hour measured in over-night polysomnography
  Interventions: Diagnostic Test: Sub-mental ultrasonography
- Moderate OSA: Patients undergoing to Sub-mental ultrasonography with Moderate sleep apnea: 15 to 29 events per hour measured in over-night polysomnography
  Interventions: Diagnostic Test: Sub-mental ultrasonography
- Severe OSA: Patients undergoing to Sub-mental ultrasonography with Severe sleep apnea: 30 or more events per hour measured in over-night polysomnography
  Interventions: Diagnostic Test: Sub-mental ultrasonography

INTERVENTIONS:
Diagnostic Test: Sub-mental ultrasonography — Sub-mental ultrasonography including tongue-base thickness, retropalatal distance and the distance between lingual arteries

SUMMARY:
The investigators hypothesize that sub-mental ultrasonography measures are strongly correlated with the severity of Obstructive Sleep Apnea Syndrome and the related specific subjective scales.

DETAILED DESCRIPTION:
Polysomnography (PSG) is the gold-standard diagnose tool for Obstructive Sleep Apnea (OSA). However, the availability of PSG is limited, particularly in developing and / or least developed countries. Sub-mental ultrasonography is stepped forward with its practical and cheap nature and its widespread use.

The investigators aimed to perform sub-mental ultrasonography to the patients who underwent to PSG by a blind-to-the-PSG-results radiologist and analyse the correlation between ultrasound measures, Apnea-Hypopnea Index (measured by Polysomnography) and subjective OSA scales.

ELIGIBILITY:
Inclusion Criteria:

* Patient who consented for sub-mental ultrasound

Exclusion Criteria:

* Any pharyngo laryngeal anatomic abnormality
* Previous history of Obstructive sleep apnea treatment
* Previous history of surgical intervention to the pharyngo laryngeal anatomic area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * For study group: Patients who have been diagnosed as having obstructive sleep apnea on polysomnography
  * For control group: Patients who have a negative polysomnography or normal scores from subjective scales
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2021-01-24 (Actual)

PRIMARY OUTCOMES:
Tongue base thickness | Baseline
  The closest distance between tongue base and the skin in the sagittal plane
Retropalatal distance | Baseline
  The diameter of retropalatal space in the transverse dimension
Distance between lingual arteries | Baseline
  Distance between lingual arteries in the transverse plane

SECONDARY OUTCOMES:
Stop-Bang questionnaire | Baseline
  This questionnaire evaluates the risk of sleep apnea. Low risk of OSA: Yes to 0-2 questions Intermediate risk of OSA: Yes to 3-4 questions High risk of OSA: Yes to 5-8 questions or Yes to 2 or more of 4 STOP questions + male gender or Yes to 2 or more of 4 STOP questions + BMI > 35 kg/m2 or Yes to 2 or more of 4 STOP questions + neck circumference.
Berlin Questionnaire | Baseline
  The questionnaire consists of 3 categories related to the risk of having sleep apnea.
  Category 1 is positive if the total score is 2 or more points. Category 2 is positive if the total score is 2 or more points. Category 3 is positive if the answer to item 10 is 'Yes' or if the BMI of the patient is greater than 30kg/m2. (BMI is defined as weight (kg) divided by height (m) squared, i.e.., kg/m2). Patients can be classified into High Risk or Low Risk based on their responses to the individual items and their overall scores in the symptom categories. High Risk: if there are 2 or more categories where the score is positive. Low Risk: if there is only 1 or no categories where the score is positive. Total score is ranged between 0-3.
Pittsburgh Sleep Quality Index (PSQI) | Baseline
  The order of the PSQI items has been modified from the original order in order to fit the first 9 items (which are the only items that contribute to the total score) on a single page. Item 10, which is the second page of the scale, does not contribute to the PSQI score. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Neck circumference | Baseline
  Neck circumference was measured with the head erect and eyes facing forward, horizontally at the upper margin of the thyroid cartilage (to the nearest 0.1 cm)
The thyromental distance | Baseline
  The thyromental distance is defined as the distance from the chin (mentum) to the top of the notch of the thyroid cartilage with the head fully extended. It is measured with a ruler

CONTACTS AND LOCATIONS:
Overall Officials: Ozge Yagcioglu Yassa, M.D., Principal Investigator — Coordinator of Sleep Disorders Centre of Bartin State Hospital
Locations (1):
- Bartin State Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shu CC, Lee P, Lin JW, Huang CT, Chang YC, Yu CJ, Wang HC. The use of sub-mental ultrasonography for identifying patients with severe obstructive sleep apnea. PLoS One. 2013 May 10;8(5):e62848. doi: 10.1371/journal.pone.0062848. Print 2013. PMID 23675433